CLINICAL TRIAL: NCT02839044
Title: A Randomized, Placebo-controlled, Double Blind Trial to Investigate Whether Vitamin K2 Can Influence Arterial Calcification in Patients With Type 2 Diabetes
Acronym: Vitacal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Yvonne T. van der Schouw, Prof., UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15/571
Record Dates: First submitted 2016-07-18; First posted 2016-07-20 (Estimated); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: Arterial Calcification; Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — menaquinone 7

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin K (Experimental): One group receives tablets of 360 microgram menaquinone-7 daily
  Interventions: Dietary Supplement: Menaquinone-7
- Placebo (Placebo Comparator): One group receives placebo tablets daily
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Menaquinone-7
  Arms: Vitamin K
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
Arterial calcification is an independent predictor of coronary events associated with a 3-4 fold increased risk of cardiovascular events. Currently, no effective intervention exists to reduce arterial calcification. However, recent studies showed that vitamin K may reduce ongoing calcium deposition in the arteries, and thereby inhibit arterial calcification.

The primary objective is to determine if MK-7 supplementation leads to stabilization or attenuation of ongoing calcium deposition in the femoral artery as quantified by 18F-NaF PET/CT imaging in patients with type 2 diabetes and arterial disease.

ELIGIBILITY:
Inclusion Criteria:

* Middle aged men and women, ≥ 40 years.
* Diagnosed with type 2 diabetes.
* Presence of arterial diseases, based on an Ankle Brachial Index (ABI) <0.9 and/or diagnosed with arterial diseases by physician.
* ABI<0.9
* Written informed consent.

Exclusion Criteria:

* Subjects participate in another intervention research or study using imaging.
* Contra-indication for undergoing18F-NaF PET/CT scan (claustrophobia, pregnancy, breastfeeding).
* Subject underwent amputation of the lower extremities (above the knee).
* Using vitamin K antagonists.
* Known coagulation problems (history of Venous Thrombo Embolism).
* Using vitamin supplements that contain vitamin K, or unwilling to stop two weeks before randomisation.
* A mean vitamin K2 intake ≥120 microgram/day measured with a questionnaire.
* Natto or goose liver consumers.
* Low kidney function (eGFR<30).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Absolute change in ongoing calcium deposition quantified as volumetric bone metabolic rate (CSUVMEAN x cm3) in the femoral artery between baseline and 6 months after baseline, as determined by 18F-NaF PET/CT imaging. | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- UMC Utrecht, Utrecht, Netherlands

REFERENCES:
- [Background] Zwakenberg SR, de Jong PA, Bartstra JW, van Asperen R, Westerink J, de Valk H, Slart RHJA, Luurtsema G, Wolterink JM, de Borst GJ, van Herwaarden JA, van de Ree MA, Schurgers LJ, van der Schouw YT, Beulens JWJ. The effect of menaquinone-7 supplementation on vascular calcification in patients with diabetes: a randomized, double-blind, placebo-controlled trial. Am J Clin Nutr. 2019 Oct 1;110(4):883-890. doi: 10.1093/ajcn/nqz147. PMID 31387121
- [Derived] Bartstra JW, Draaisma F, Zwakenberg SR, Lessmann N, Wolterink JM, van der Schouw YT, de Jong PA, Beulens JWJ. Six months vitamin K treatment does not affect systemic arterial calcification or bone mineral density in diabetes mellitus 2. Eur J Nutr. 2021 Apr;60(3):1691-1699. doi: 10.1007/s00394-020-02412-z. Epub 2020 Oct 17. PMID 33068157